CLINICAL TRIAL: NCT05932420
Title: Role of Intermittent Exogenous Ketosis in the Physiological and Muscular Adaptive Response to Endurance Training. A Study in Young, Male Volunteers.
Brief Title: Role of Intermittent Exogenous Ketosis in the Physiological and Muscular Adaptive Response to Endurance Training
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Ruben Robberechts, Mr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: S66150
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Exercise Adaptations
Keywords: ketone bodies; Exercise adaptations; Sleep
MeSH Terms: interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Placebo is provided
  Interventions: Dietary Supplement: Placebo
- Experimental groep (Experimental): Ketone ester is provided
  Interventions: Dietary Supplement: Ketone ester

INTERVENTIONS:
Dietary Supplement: Placebo — 16.4g pure medium triglyceride oil mixed with 1 mM of bitter sucrose octaacetate. A dose of 25g of the placebo drink is provided immediately after each training session and 30 minutes before sleeptime throughout the training period.
  Arms: Control group
Dietary Supplement: Ketone ester — A dose of 25g of ketone ester after each training session and 30 minutes before sleeptime throughout the training period.
  Arms: Experimental groep

SUMMARY:
In a recent study (Poffé et al., 2019), we demonstrated that increasing the concentration of ketone bodies in the blood through the ingestion of a ketone ester (KE) post-exercise and just before sleeping time during a 3-week overtraining period resulted in suppression of the physiological symptoms of overtraining. Consistent KE intake improved endurance performance, positively affected the autonomic regulation of the heart, suppressed the increase of nocturnal sympathetic activity, and increased spontaneous energy intake. In addition, KE intake had a positive effect on muscular adaptive response, as evidenced by the significantly increased muscular angiogenesis. Therefore, in this study, we aim to investigate whether the oral administration of ketones after exercise and just before bedtime also has a positive effect on the adaptive response during a well-dosed endurance training program. Since suppression of nocturnal sympathetic activity can positively influence sleep quality, we will also study the effect of KE and the training period on sleep quality.

To investigate this, we will use a randomized, placebo-controlled parallel research design. Well-trained male cyclists will participate in a fully controlled intervention period of 8 weeks. During the intervention period, participants will follow a supervised cycling training program (5-7 training sessions per week) with a gradual buildup aimed at improving endurance capacity.

Throughout the intervention period, participants will ingest 25g ketone ester or a corresponding placebo after each training session and 30 minutes before bedtime. Endurance performance will be evaluated before the start of the training period (pretest), after week 3 (midtest), after week 7 (posttest) of the training period, and at the end of the training intervention (posttest+taper). Additionally, blood samples will be taken at the pre-test and post-test to analyze markers of hormonal status and inflammation. Muscle biopsies will be taken from the vastus lateralis muscle of the right leg at pretest and posttest to analyze cross-sectional area, muscle fiber typing, angiogenesis, protein synthesis and degradation, mitochondrial function, and energy substrate concentrations. One month after the intervention period, an additional biopsy will be taken to study changes in gene expression (epigenetic modifications). Sleep will be evaluated via polysomnography (PSG) at the pretest, midtest and posttest. Finally, before and after the training period, resting and exercise echocardiography will be taken to investigate investigate structural and morphological changes of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Physically fit and regularly involved in physical activity (2-5 exercise sessions of > 30min per week)
* Good health status confirmed by a medical screening
* VO2max higher than 50 ml.min-1.kg-1
* Body Mass Index (BMI) between 18 and 25
* Normal sleep pattern as assessed by the Pittsburgh Sleep Quality Index (PSQI, appendix 2)

Exclusion Criteria:

* Any kind of injury/pathology that is a contra-indication to perform high-intensity exercise
* Intake of any medication or nutritional supplement that is known to affect exercise performance or sleep
* Intake of analgesics, anti-inflammatory agents, or supplementary anti-oxidants, from 2 weeks prior to the start of the study.
* Night-shifts or travel across time zones in the month preceding the study
* Blood donation within 3 months prior to the start of the study
* Smoking
* More than 3 alcoholic beverages per day or more than one glass if wine per day
* Involvement in elite athletic training at a semi-professional or professional level
* Any other argument to believe that the subject is unlikely to successfully complete the full study protocol

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean power output during a 30min cycling time trial | Pretest (before the start of the training intervention) - Midtest (after week 3 of the training intervention) - Posttest (after week 7 of the training intervention) - Posttest+taper (after week 8 of the training intervention)
  Change in mean power output during a self-paced 30 min cycling time trial on a cyling ergometer
Change in capillarization of the musculus vastus lateralis | Pretest (before the start of the training intervention) - Posttest (after week 7 of the training intervention)
  Change in capillarization (CFPE-index) of the musculus vastus lateralis
Change in sleep efficiency | Pretest (before the start of the training intervention) - Midtest (after week 3 of the training intervention) - Posttest (after week 7 of the training intervention)
  Change in sleep efficiency measured by polysomnography
Change in REM sleep | Pretest (before the start of the training intervention) - Midtest (after week 3 of the training intervention) - Posttest (after week 7 of the training intervention)
  Change in REM sleep measured by polysomnography

SECONDARY OUTCOMES:
Change in the nocturnal urinary excretion of dopamine | Pretest (before the start of the training intervention) - Midtest (after week 3 of the training intervention) - Posttest (after week 7 of the training intervention)
  Change in the nocturnal urinary excretion of dopamine
Change in the nocturnal urinary excretion of noradrenaline | Pretest (before the start of the training intervention) - Midtest (after week 3 of the training intervention) - Posttest (after week 7 of the training intervention)
  Change in the nocturnal urinary excretion of noradrenaline
Change in the nocturnal urinary excretion of adrenaline | Pretest (before the start of the training intervention) - Midtest (after week 3 of the training intervention) - Posttest (after week 7 of the training intervention)
  Change in the nocturnal urinary excretion of adrenaline
Change in maximal oxygen uptake | Pretest (before the start of the training intervention) - Midtest (after week 3 of the training intervention) - Posttest (after week 7 of the training intervention)
  Change in maximal oxygen uptake measured during a maximal incremental exercise test on a cycling ergometer

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Research Group, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Poffe C, Ramaekers M, Van Thienen R, Hespel P. Ketone ester supplementation blunts overreaching symptoms during endurance training overload. J Physiol. 2019 Jun;597(12):3009-3027. doi: 10.1113/JP277831. Epub 2019 May 22. PMID 31039280
- [Background] Robberechts R, Albouy G, Hespel P, Poffe C. Exogenous Ketosis Improves Sleep Efficiency and Counteracts the Decline in REM Sleep after Strenuous Exercise. Med Sci Sports Exerc. 2023 Nov 1;55(11):2064-2074. doi: 10.1249/MSS.0000000000003231. Epub 2023 Jun 1. PMID 37259248